CLINICAL TRIAL: NCT03949764
Title: Increasing Access to Hepatitis C Treatment in Opioid Endemic Rural Areas: The Kentucky Viral Hepatitis Treatment (KeY Treat) Study
Brief Title: The Kentucky Viral Hepatitis Treatment Study
Acronym: KeY Treat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jennifer Havens (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH); Gilead Sciences (Industry); University of Kentucky (Other); Icahn School of Medicine at Mount Sinai (Other); University of Bristol (Other)
Responsible Party: Sponsor-Investigator, Jennifer Havens, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47239; R01DA047952 (NIH)
Record Dates: First submitted 2019-05-02; First posted 2019-05-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis C; Opioid-Related Disorders; Injection Drug Use
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders | interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HCV Positive Study Participants (Experimental): Study participants will be administered a standard 12-week course of sofosbuvir/velpatasvir (Epclusa®).
  Interventions: Drug: Sofosbuvir/velpatasvir (Epclusa®)
- Control (Pike County) (No Intervention): After completion of the study, we will compare HCV incidence and prevalence rates in Perry County (intervention) and Pike County (control). This will be measured through data provided by the local health departments of each county. Confidential Hepatitis C screening will be conducted in some cases, and resources will be provided to those testing positive but they will not receive treatment as part of this study.

INTERVENTIONS:
Drug: Sofosbuvir/velpatasvir (Epclusa®) — The protocol is intended to follow best practices/standard of care for the treatment of HCV, with additional allowances for the investigators to apply rigorous scientific practices for the research aspects of the study. While the treatment of HCV is fairly straightforward, less is known about treating active drug users and RNA-positive individuals in rural areas. We propose eight visits, including intake, four treatment-related visits, and three visits to determine re-infection (6- and 12-months post-SVR). Because determination of medication adherence and long-term reinfection rates are not part of standard clinical practice, the rural protocol developed at the conclusion of KeY Treat will be streamlined based on findings, consisting of five or fewer clinical contacts. The drug used for treatment is Epclusa®, a 12-week, once per day, pan-genotypic DAA with a favorable side effect profile. Vosevi® will also be available in cases where participants are non-responsive or are re-infected.
  Arms: HCV Positive Study Participants

SUMMARY:
The overarching goal of the Kentucky Viral Hepatitis Treatment Project (KeY Treat) is to increase hepatitis C virus (HCV) treatment access and delivery in a rural Appalachian community, which is in the midst of the opioid/hepatitis C (HCV) syndemic. KeY Treat is a clinical research study seeking to determine whether removing barriers (cost, insurance, specialist, abstinence) associated with accessing direct-acting antivirals (DAAs) for the treatment of HCV will impact health in Perry County, Kentucky.

DETAILED DESCRIPTION:
The overarching goal of the Kentucky Viral Hepatitis Treatment Project (KeY Treat) is to increase access to treatment for the hepatitis C virus (HCV) in a rural Appalachian community in the midst of the opioid/HCV syndemic. This study seeks to examine whether removing barriers associated with accessing direct-acting antivirals (DAAs) for the treatment of HCV (high out-of-pocket costs, insurance restrictions requiring a specialist, abstinence, and significant liver damage) will significantly reduce the burden of HCV in Perry County, Kentucky. The proposed study is made possible by a significant drug donation from Gilead Sciences for sofosbuvir/velpatasvir, a 12-week, once per day, pan-genotypic DAA. KeY Treat proposes a multi-pronged approach to treating HCV using a mid-level provider model. In addition to DAA treatment, participants will be offered access to subsidized medication-assisted treatment, syringe services, and case management. Existing resources in the target community (public health, jail, hospital) will be leveraged, as well as ongoing projects dedicated to increasing access to HCV care in affected communities (ECHO, FOCUS) to answer whether removing the major barriers to HCV treatment affect access, and what barriers remain. All RNA-positive residents of Perry County, Kentucky will be eligible/recruited for study participation (N≈900), and the following specific aims will be addressed: 1) determination of HCV treatment uptake among rural residents with chronic HCV; 2) examination of the predictors of treatment completion among those enrolled in KeY Treat; 3) examination of the characteristics of participants achieving sustained virologic response (SVR, or cure); 4) establishment of long-term re-infection rates among those achieving SVR; 5) examination of 5-year reductions in incidence and prevalence of HCV in the intervention community compared with a control county in rural Kentucky; and 6) evaluate the impact and cost-effectiveness of KeY Treat using mathematical modeling. The proposed research has tremendous potential to impact public health in the rural United States. The majority of counties identified in CDC's recent HCV/HIV hotspot analysis were rural, and there is a real need to improve access to DAAs in order to prevent further HCV transmission, reduce the burden of advanced liver disease, and hepatocellular carcinoma in generations to come. Data from KeY Treat will inform policies around Medicaid/insurance restrictions for DAAs, and will deliver a much needed blueprint for the provision of HCV treatment in resource-deprived rural areas.

ELIGIBILITY:
Inclusion Criteria:

* RNA positive for HCV
* Perry County residency (verified via ID card showing local address, lease, utility bill, etc.)
* 18 years of age or older

Exclusion Criteria:

* Individuals who are unable to provide consent (to be determined by local study staff in conjunction with our psychiatrist, Dr. Lofwall, a Co-I on the study)
* Individuals under 18 years of age (study drugs not FDA-approved for those <18)
* Pregnant women (unable to participate during duration of pregnancy, but encouraged to return following delivery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment Uptake | Visits 1-5, 1 to 12 weeks post-baseline
  Defined as receiving the first dose of medication, to be measured by number of pills left and viral load.
Treatment Completion | Visit 6, 24 weeks post-baseline
  Defined as receiving all doses of medication, to be measured by number of pills left and viral load.
Sustained Virologic Response (SVR) | Visit 7, 50 weeks post-baseline
  Defined as undetectable viral RNA at the 12-week post-completion blood draw (SVR-12).
Re-infection | Visit 8, 102 weeks post-baseline
  Defined as the presence of viral RNA at either the 6- or 12-month follow-up after achieving SVR.

SECONDARY OUTCOMES:
Prevalence of HCV | Visit 8, 102 weeks post-baseline
  Prevalence of HCV in study population, measured by viral load.
Incidence of HCV | Visit 8, 102 weeks post-baseline
  Incidence of HCV in study population, measured by viral load and new cases.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Havens, PhD, Principal Investigator — University of Kentucky Ctr on Drug & Alcohol Rsrch
Locations (1):
- ARH Medical Mall, Hazard, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Havens JR, Schaninger T, Fraser H, Lofwall M, Staton M, Young AM, Hoven A, Walsh SL, Vickerman P. Eliminating hepatitis C in a rural Appalachian county: protocol for the Kentucky Viral Hepatitis Treatment Study (KeY Treat), a phase IV, single-arm, open-label trial of sofosbuvir/velpatasvir for the treatment of hepatitis C. BMJ Open. 2021 Jul 5;11(7):e041490. doi: 10.1136/bmjopen-2020-041490. PMID 34226208

DOCUMENTS (1):
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT03949764/ICF_000.pdf